CLINICAL TRIAL: NCT06975228
Title: TReating Unhelpful Suspicious Thoughts in Adolescents (TRUST): a School-based Case Series
Acronym: TRUST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 191567
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Paranoia
Keywords: Paranoia; Adolescents; School; Feasibility; Acceptability
MeSH Terms: conditions — Paranoid Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRUST (Experimental): Six session psychological intervention focussing on imagery and values
  Interventions: Behavioral: TRUST

INTERVENTIONS:
Behavioral: TRUST — Six-session psychological intervention focussing on values and imagery Session 1: Assessment, formulation and psychoeducation Session 2: Values and values-based goals Session 3-5: Harnessing imagery to pursue values and imagery focussed strategies to change negative beliefs about self and others Session 6: Review

SUMMARY:
The goal of this acceptability and feasibility trial is to identify whether a six-session intervention for suspicious thoughts is feasible and acceptable to school-based adolescents.

The main research question is:

Is it feasible and acceptable to offer a brief imagery and values-based intervention for adolescents experiencing paranoia in schools?

Aims The primary aim of the current study is to identify whether a six-session brief intervention delivered in schools is feasible and acceptable to young people experiencing paranoia. Secondarily, it aims to identify preliminary outcomes of such an intervention on levels of paranoia, as measured by the Revised Green et al., Paranoid Thoughts Scale (R-GPTS).

Participants will be screened for paranoid thoughts and those eligible will be offered a six-session intervention. Participants will be asked to complete various measures prior to and following therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 16+
* Attending participating school
* Low risk
* No current mental health support
* Symptoms of paranoia i.e. scoring above 11 on R-GPTS part B subscales, equating to "moderately severe" paranoia and above

Exclusion Criteria:

* evidence of a primary alcohol or substance dependence issue at initial assessment;
* developmental disability;
* not fluent in English (due to questionnaire validity issues);
* receiving another therapy at the same time;
* moderate to high levels of risk

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Throughout course of study - 18 months
  GREEN: > 5 participants of target recruited AMBER = 3 to 4 of target recruited RED < 2 of target recruited
Retention | Throughout course of study - 18 months
  GREEN: 5 or more of participants providing end of therapy assessment outcome data AMBER: 3 to 4 participants providing end of therapy assessment outcome data RED: 2 or less of participants providing end of therapy assessment outcome data
Adherance | Throughout course of study - 18 months
  GREEN= 5 or more participants attend at least 3 sessions of therapy AMBER>= 3 to 4 participants attend at least 3 sessions of therapy RED: 2 or less of participants attend at least 3 sessions of therapy
Acceptability | End of patient involvement
  Acceptability of the therapy will be assessed via therapy process feedback questionnaire given to participants upon therapy completion or withdrawal and adverse effects of study participation questionnaire.

SECONDARY OUTCOMES:
Revised Green et al., Paranoid Thoughts Scale (R-GPTS) Part B | Weekly sessions
  For screening of and assessing adolescents' paranoia, Revised Green et al., Paranoid Thoughts Scale (R-GPTS) will be used due to high reliability. The R-GPTS comprises of two subscales assessing for frequency of ideas of references (eight questions) and ideas of persecution (10 questions) on a five-point Likert scale. Part B will be used. "The R-GPTS score ranges are: average (Reference: 0-9; Persecution: 0-4); elevated (Reference: 10-15; Persecution: 5-10); moderately severe (Reference: 16-20; Persecution:11-17); severe (Reference: 21-24; Persecution: 18-27); and very severe (Reference: 25+; Persecution: 28+)". Clinical cut-offs on the persecution scales are 11 for persecutory ideation. Higher levels of RGPTs scores indicate higher difficulties.
Comprehensive Assessment of Acceptance and Commitment Therapy processes for Youth (compACT-Y; Morey et al., 2024) | Baseline assessment, post-therapy (following six sessions), 6 week follow-up
  The compACT-Y consists of 19-items scored on a six-point likert scale to assess psychological flexibility, with higher scores indicating higher flexibility. This includes the three factors of valued action, openness to experience and behavioural awareness, all linking to acceptance and commitment therapy (ACT) frameworks and methodology. This has been identified to be a valid and reliable measure for the use in young people.
Negative mental imagery questionnaire (MIQ-N) | Baseline assessment, post-therapy (following six sessions), 6 week follow-up
  The MIQ-N consists of 16-items assessing for experiences of mental images. It has four sub-scales: intrusiveness, realness, controllability and beliefs about mental imagery. Participants are asked to rate how true each of the statements are to them on a seven-point Likert scale. Cronbach's alpha ranges from 0.84 - 0.90 when each of the subscales have been tested for reliability. The higher the score the higher the experience of negative mental images.
Brief Core Schema Scale (BCSS) | Baseline assessment, post-therapy (following six sessions), 6 week follow-up
  The BCSS evaluates self and other beliefs using a 24-item scale, rating positive and negative self and other beliefs. Participants are asked to initially rate whether they hold the belief on yes/no and then rate the strength of the belief using a four-point Likert scale. Negative evaluations of self and others are suggested to be indicative of paranoia in the general population. The measure has good internal consistency for non-clinical samples (α = 0.74) and good retest-reliability for all subscales.
Work and Social Adjustment Scale - Youth (WSAS-Y) | Baseline assessment, post-therapy (following six sessions), 6 week follow-up
  The WSAS-Y is a measure of functionality for young people in areas such as school, relationships and activities. It has five subscales and assesses severity of impairment using an eight-point scale, generating a total score out of 40, with greater scores indicating greater impairment. It has been suggested to have high internal consistency (α = 0.84) and reliability (r = 0.80).
Imagery characteristics | Baseline assessment, post-therapy (following six sessions), 6 week follow-up
  The weekly imagery characteristics scale is a seven-item measure rating the characteristics of mental images including how real or pre-occupying they are. Participants are asked to rate each item on a 10-point scale from 'not at all' to 'extremely'.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanson School, Bradford, United Kingdom